CLINICAL TRIAL: NCT01623440
Title: Neural Correlates of Food Reward in Native American Women
Brief Title: Food Reward in Native American Women
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 10152
Record Dates: First submitted 2012-06-12; First posted 2012-06-20 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Naltrexone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Placebo/Naltrexone and fMRI: A placebo or Naltrexone will be given before fMRI. All participants will undergo both procedures. Naltrexone/placebo are not used as an intervention.
  Interventions: Combination Product: Placebo and fMRI; Combination Product: Naltrexone and fMRI

INTERVENTIONS:
Combination Product: Placebo and fMRI — Pill form, participant dosed one time an hour before fMRI.
Combination Product: Naltrexone and fMRI — 50 mg pill given one time, one hour before fMRI

SUMMARY:
This study aims to characterize the neurobiology of obesity in American Indians (AI) using functional MRIs to examine the correlation between brain response to food stimuli in AI women. A functional MRI (fMRI) is used to visualize brain activity when obese and lean AI women look at images of fattening food, non-fattening food and non-food objects. Additionally examined is the effect of the drug naltrexone to suppress brain response to visual food cues and calorie intake in the women.

DETAILED DESCRIPTION:
The study looks at both obese and lean women. Each woman comes in for two visits. Each woman takes both the Naltrexone or placebo (one during each visit). Research staff and participants are blinded. Drugs are not used as treatment, but rather to provide information for possible future treatments.

Hypotheses are:

1. Compared with their lean counterparts, obese women will demonstrate more fMRI activation in the brain in response to visual food cues.
2. Naltrexone will reduce the activation in reward-relevant brain sites in response to viewing photographs of fattening food as compared in placebo in both groups.
3. Naltrexone will suppress spontaneous intake of food in obese and lean AI women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Self-identified AI
* BMI over 30 OR between 20 and 24.9
* Must see clearly with or without glasses
* Capable of giving informed consent

Exclusion Criteria:

* Smokes more than one cigarette a day
* Drinks more than two alcoholic drinks a day
* Uses recreational drugs
* Is pregnant
* Has had weight loss surgery
* Other major medical problems (e.g. diabetes)
* Taking medications that alter appetite or body weight
* Significant food allergies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females Only
Study Population: Self-identified Native American women between ages of 18 and 45.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
fMRI activation in the brain in response to visual food cue | With In 30days
  fMRI activation in the brain in response to visual food cue

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Beckman, MD, MPH, Principal Investigator — Division of Endocrinology, Diabetes & Metabolism, University of Minnesota Department of Medicine
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No